CLINICAL TRIAL: NCT02138292
Title: A Phase 1B Clinical Trial of Trametinib Plus Digoxin in Patients With Unresectable or Metastatic BRAF Wild-type Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 012014-007
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — trametinib; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trametinib (2mg)/Digoxin (0.25mg) (Experimental): 1. Trametinib (2mg) will be administered orally on a daily basis.
  2. Digoxin (0.25mg) will be administered orally on a daily basis.
  On a 8-week cycle, duration of treatment can last from 8 to 104 weeks.
  Interventions: Drug: Trametinib (2mg)/Digoxin (.25mg)

INTERVENTIONS:
Drug: Trametinib (2mg)/Digoxin (.25mg) — 1. Trametinib (2mg) will be administered orally on a daily basis.
  2. Digoxin (0.25mg) will be administered orally on a daily basis.
  On a 8 week cycle, duration of treatment can last from 8 to 104 weeks.

SUMMARY:
The study is a prospective, single-arm, one-site therapeutic trial of the combination of trametinib plus digoxin for advanced melanoma. endpoints are toxicities assessed by nCi CTCae v4.1 within the first 8 weeks, responses measured by ReCiST v1.1 criteria every 8 weeks with scans and exams, tumor sensitivity to the drug combination quantified by tumor regressions in nSG mice, and correlations of response with tumor sensitivity, BRaF status, MaPK inhibitor exposure history, and tumor sodium pump expression.

Treatment Dosage and administration

Study Drugs:

1. Trametinib (2mg) will be administered orally on a daily basis.
2. Digoxin (0.25mg) will be administered orally on a daily basis.

on a 8-week cycle, duration of treatment can last from 8 to 104 weeks.

endpoints

1. Toxicities will be assessed via nCi's CTCae v4.1 toxicity criteria. DLTs will be defined based on the rate of drug-related (definitely or probably) grade 3-5 adverse events experienced within the first 8 weeks of study treatment. The MTD will be exceeded if more than 20% of patients on the study experience DLTs.
2. Responses will be measured by ReCiST v1.1 every 8 weeks. Response duration will be defined as time from first documented response until disease progression. PFS is time from treatment until disease progression.
3. Patient tumor sensitivity to the drug combination will be quantified by the amount of subcutaneous established tumor growth inhibition in nSG mice by 5d/week oral gavage with drugs.
4. Tumor nRaS status will be determined by tumor Dna extraction, PCR amplification of exons and Sanger sequencing of nRaS.
5. History of prior MaPK inhibitor therapies will document MeK inhibitor exposures.
6. Sodium pump subunit expression will be analyzed by pretreatment tumor immunohistochemistry and a qualitative 0 to 3+ grading system.

DETAILED DESCRIPTION:
Primary Objectives:

* To describe the toxicities and estimate the frequency of dose limiting toxicities (DLTs) of digoxin in combination with trametinib in advanced melanoma patients and estimate the frequency of DLTs.
* To measure the response rate, response duration and progression free survival (PFS) of digoxin plus trametinib in advanced melanoma.

Secondary Objectives:

* To correlate NSG xenograft sensivity to the drug combination with clinical response in the same patient.
* To compare response rates in MAPK inhibitor naive versus refractory patients and NRAS mutant versus wild-type patients and for sodium pump 3 subunit high tumor expression versus low tumor expression patients.

Rationale: Having established cell culture and xenograft systems for studying patient melanoma samples, the researchers were able to grow tumors in vitro and in vivo from single cells and found a correlation of tumor metastatic behavior in immunocompromised mice and in patients. Recently they have extended the experiments to examine melanoma sensitivity to novel compounds. In screens of FDA approved drugs, they found several cardenolides including digoxin that reproducibly exhibited greater toxicity to primary human melanomas as compared to a range of normal human cells. They then examined the anti-tumor efficacy against primary human melanomas growing in vivo as xenografts. While trametinib, vemurafenib, and digoxin and digitoxin individually slowed the growth of human melanomas xenografts, they did not cause tumor regression. However, the combination of digoxin or digitoxin and trametinib caused substantial tumor regression using melanomas obtained from multiple patients, some with BRAF mutations and some without. The effects were dramatically better than trametinib, digoxin, digitoxin or vemurafenib alone. No difference in efficacy for the combination was seen in BRAF mutant and BRAF wild-type samples.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologic diagnosis of unresectable or metastatic melanoma. For unknown primary disease, diagnosis of metastatic disease by cytology FNA is not acceptable. BRAF wild-type confirmed, and NRAS mutation assessed.

  2. Age > 18 years.

  3. Any number of prior systemic therapeutic regimens for unresectable stage III or stage IV melanoma. This includes chemotherapy, immunotherapy, pathway inhibitors, biochemotherapy, or investigational treatments. Patients may also have received therapies in the adjuvant setting.

  4. ECOG Performance status 0-2.

  5. Adequate organ and marrow function as defined below:
* leukocytes ≥ 2,000/mcL
* absolute neutrophil count ≥ 1,000/mcL
* platelets ≥ 75,000/mcl
* total bilirubin < 3 x institutional upper limit of normal
* AST(SGOT)/ALT(SPGT) ≤ 2.5 X institutional upper limit of normal
* creatinine < 1.5 mg/dL
* cardiac ejection fraction > 50%
* QTc < 480msec

  6. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria: Has not undergone a hysterectomy or bilateral oophorectomy; or Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

  7. All sites of disease must be evaluated within 4 weeks prior to beginning therapy. Patients must have measurable disease as defined by RECIST v1.1.

  8. Ability to understand and the willingness to sign a written informed consent.

  9. Patients must be willing to undergo tumor biopsy pretreatment and at relapse.

Exclusion Criteria:

1. Subjects who have had chemotherapy or radiotherapy or any systemic therapy for melanoma within 2 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier. No concomitant therapy is allowed including IL2, interferon, ipilimumab, anti-PD-1 or anti-PD-L1 antibody, cytotoxic chemotherapy, immunosuppressive agents, or other investigational therapies.
2. Active infection with hepatitis B or C or HIV.
3. Subjects with active CNS disease are excluded. Patient with brain metastases previously treated with surgery or radiation therapy and with confirmed SD for >4 weeks are allowed.
4. Patients are excluded if they have a history of any other malignancy from which the patient has been disease-free for less than 2 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix.
5. Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Cardiac symptoms or events within 24 weeks.
6. History of predisposition to retinal vein occlusion or central serous retinopathy.
7. Inability to assess BRAF or NRAS mutation status. Hypersensitivity to digoxin.
8. Wolff-Parkinson White syndrome or AV block or sinus node dysfunction.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-07; Primary Completion 2017-02-23 (Actual); Study Completion 2017-02-23 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Doxicities (DLTs) | within the first 8 weeks of study treatment
  To describe the toxicities and estimate the frequency of dose limiting toxicities (DLTs) of digoxin in combination with trametinib in advanced melanoma patients and estimate the frequency of DLTs.

SECONDARY OUTCOMES:
Response Rate | up to 104 weeks
  Responses will be measured by RECIST v1.1 every 8 weeks. Response duration will be defined as time from first documented response until disease progression. PFS is time from treatment until disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Frankel, MD, Principal Investigator — Professor Internal Medicine-Hematology Oncology
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States